CLINICAL TRIAL: NCT04519723
Title: Laser 360iQ: Optimal Light-laser Combination Therapy for the Improvement of Skin Color, Tone, Texture and Laxity.
Brief Title: Laser 360iQ: Optimal Light-laser Combination Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Lasers Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYZ-12345-2012
Record Dates: First submitted 2014-01-07; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2012-04

CONDITIONS: Photodamage
Keywords: Hyperpigmentation; telangiectasias
MeSH Terms: conditions — Hyperpigmentation; Telangiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alma Harmony Laser System (Other): There is only one arm. Three hand modules; Dye-VL 500-600nm, High Power QSW 1064nm, and High power Pixel ER:YAG 2940nm laser module with rollers will be utilized in combination in a series of treatments intended to improve skin color, tone, texture and laxity. Subjects will receive up to four treatments administered in intervals of 28 +/- 2 days. Treatment duration of approximately 60 minutes.
  Interventions: Device: Assess the safety and efficacy of light-laser therapy using the Harmony XL and Dye-VL (500-600nm), Q-Switched 1064nm, Er:YAG 2940nm modules in combination .

INTERVENTIONS:
Device: Assess the safety and efficacy of light-laser therapy using the Harmony XL and Dye-VL (500-600nm), Q-Switched 1064nm, Er:YAG 2940nm modules in combination .

SUMMARY:
To assess the safety and efficacy of light-laser combination therapy for the improvement of skin color, tone, texture and laxity

DETAILED DESCRIPTION:
This is a prospective study to test the safety and efficacy of a three different light and laser handpieces for the improvement of skin color, tone, texture and laxity. All subjects will receive up to four treatments, administered in intervals of 28 +/- 2 days. Each full face treatment duration will be approximately 60 minutes. The initial power and number of passes parameters shall be set according to the clinical indication and skin type of the subject treated. The treatment area will be cleaned and photographed before each treatment. Photographs will be taken at baseline, prior to each treatment and during each follow-up visit. Before the initiation of the first treatment each subject will undergo clinical evaluation.

Clinical improvement will be assessed by the investigator from the visual appearance of the treated area and from the fixed magnification clinical photographs according to the following scale: -1 for exacerbation, 0 no change, 1 for 1%-25% improvement, 2 for 25%-50% improvement, 3 for 50%-75% improvement, and 4 for 75%-99% improvement. Adverse side effects will be scored by clinical evaluation of erythema, edema, and burns. Treatments and results will be documented in a Case Report Form at each treatment session and follow-up session (1 month and 3 months after the last treatment). In case of adverse side effects and symptoms other than erythema or edema appear during or following a treatment, the next treatment may be skipped by two weeks or treatment parameters reduced until symptoms resolve. If adverse side effects are observed, the investigator should provide the subject with the proper care and remedy and will document it in the Case Report Form.

ELIGIBILITY:
Inclusion Criteria:

* Male or female in good general health between 35 to 60 years of age.
* Must be willing to execute informed consent. Patient must also consent to having photos taken at each visit.
* A potential subject must exhibit:

Facial wrinkling and graded mild to moderate overall rough texture, large pores, and/or skin laxity.

* For FEMALE PATIENTS OF CHILDBEARING POTENTIAL, must have had a regular menstrual cycle prior to study entry (a female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation) and is willing to use an acceptable form of birth control during the entire course of the study [i.e., acceptable methods of birth control are oral contraceptives, contraceptive patches/rings/implants Norplanit®, Depo-Provena®, double-barrier methods (e.g. condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control should the subject become sexually active]. All systemic birth control measures must be in consistent use at least 30 days prior to study participation.
* Negative urine pregnancy test results at the time of study entry (if applicable).
* Must be willing to comply with study visits and complete the entire course of the study.

Exclusion Criteria:

* Negative urine pregnancy test results at the time of study entry (if applicable).
* Must be willing to comply with study visits and complete the entire course of the study.

Subjects meeting any of the following criteria will be excluded from participation:

The following are exclusion criteria for subjects in this study:

* A subject with any UNCONTROLLED systemic disease. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
* A subject with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
* A subject using any topical product containing a retinoid, retinol, or other vitamin A derivative within 3 months prior to or during the study period.
* A subject using any systemic steroid therapy within 6 months prior to or during the study period.
* A subject that has been treated with Botox/Dysport or filler/biostimulatory molecule injections to his/her face within the past six months.
* A subject using any topical medicated creams, lotions, powders, etc. on the treatment areas during the study period, other than the study treatment regimen within 14 days.
* A subject that has previously been treated with systemic retinoids within the past year (e.g., Accutane®, Roche Dermatologics).
* A subject with recently excessive facial exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing). During the study, when excessive sun exposure is unavoidable, subjects must wear appropriate protective clothing (e.g. hat) and comply with the study dosing regimen of daily application of the dispersed sunblock.
* A subject with a recent history or active presence of any facial skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e. moderate to severe acne vulgaris, atopic dermatitis, psoriasis, rosacea, seborrheic dermatitis, excessive facial hair or coloration).
* A female subject who is pregnant, nursing an infant or planning a pregnancy during the study [throughout the course of the study, women of child-bearing potential must use reliable forms of contraception (i.e., oral contraceptive, intrauterine device, abstinence, or spermicides and condoms used in combination)].
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.
* Subjects who are pregnant, breast-feeding, or planning a pregnancy. Females of childbearing potential, in addition to having a negative pregnancy test at the screening visit, must be either:

  * using the same form (i.e. brand) and dosage regimen of an oral contraceptive pill or of a hormonal implant continuously for three months prior to study entry and continue during the entire study, or
  * willing to use a different form of birth control during the study other than any form of hormonal methods such as oral contraceptive pills and hormonal implants 30 day prior to study entry and during the entire study period. For the purpose of this study, the following are considered acceptable methods of birth control: double-barrier methods (e.g.: condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control should the subject become sexually active.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Visual observation of improvement in photoaging | The investigator will evaluate the change in visual appearance of the treated area before one month, two month, and three month treatments and before each follow-up visit (1 month and 3 months after the last treatment).
  The investigator will evaluate the clinical improvement from the visual appearance of the treated area and from the fixed magnification clinical photographs according to the following Global Assessment scale (compared to baseline photographs):
  Global Aesthetic Improvement Scale (GAIS )
  Rating Description
  1. = Very much improved 75%-99%
  2. = Much improved 50%-75% 3= Improved 25%-50% 4= No change 1%-25% 5=Worse <1%

CONTACTS AND LOCATIONS:
Overall Officials: Brian Zelickson, MD, Principal Investigator — Board Certified Dermatologist
Locations (1):
- Zel Skin & Laser Specialist, Edina, Minnesota, United States